CLINICAL TRIAL: NCT01518218
Title: Effectiveness of Laying-on-of-hands for Patients With Sickle Cell Disease in Africa
Brief Title: Effectiveness of Laying-on-of-hands for Sickle Cell Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MOA Health Science Foundation (Other)
Responsible Party: Principal Investigator, Kiyoshi Suzuki, president, MOA Health Science Foundation
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MOA-002
Record Dates: First submitted 2012-01-21; First posted 2012-01-25 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2012-01

CONDITIONS: Sickle Cell Disease; Pain Crisis Recurrent; Anemia; Infection; Death
Keywords: Sickle cell disease; laying-on-of-hands; morbidity; mortality
MeSH Terms: conditions — Anemia, Sickle Cell; Anemia; Infections; Death | interventions — Therapeutic Touch

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- laying-on-of-hands (Experimental): Patients of this arm received laying-on-of-hands twice a day (45 minutes each) every weekday for 1year, and received conventional medical treatment if necessary.
  Interventions: Behavioral: laying-on-of-hands
- control group (No Intervention): Patients of this arm did not receive any alternatives other than conventional treatment.

INTERVENTIONS:
Behavioral: laying-on-of-hands — The intervention group received laying-on-of-hands every weekday for 1 year along with conventional medicine. The control group did not undergo any alternatives to OPT.
  Other Names: Okada Purifying Therapy; biofield therapy
  Arms: laying-on-of-hands

SUMMARY:
The objective of this study is to evaluate the effectiveness of 1-year administration of laying-on-of-hands on the morbidity and mortality of patients with sickle cell disease in Africa.

DETAILED DESCRIPTION:
Patients with sickle cell disease (SCD) have a high risk of premature death in Africa, mainly due to insufficient medical services. SCD patients often visit emergency department and need hospitalization when they suffer from severe pain; however, they manage most of painful episodes at home. Appropriate pain management at home is, therefore, crucial to improve their clinical course and quality of life. Laying-on-of-hands may be a good candidate for home care management, because family member(s) can become a practitioner of laying-on-of-hands without difficulty and administer it to their loved one as an initial treatment whenever necessary. There are no reports concerning the effectiveness of laying-on-of-hands for the outcomes of SCD patients, as far as we have investigated.

ELIGIBILITY:
Inclusion Criteria:

* patients with symptoms associated with sickle cell disease
* those able to receive laying-on-of-hands every weekday for 1 year
* those able to receive conventional medical treatment whenever necessary
* those able to receive blood test at the beginning, after 6 month and after 1 year

Exclusion Criteria:

* those who wish to use other complementary and alternative therapies along with laying-on-of-hands

Ages: 3 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2006-03; Primary Completion 2007-03 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
disease-related episodes and mortality | 3 years and 9 months

SECONDARY OUTCOMES:
blood data | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kodondi K Koto, MD, PhD, Study Director — The Institute of Scientific Research for Health, Kinshasa
Locations (1):
- The national medical center for sickle cell disease, Kinshasa, Democratic Republic of the Congo

REFERENCES:
- [Derived] Minga TM, Koto FK, Egboki H, Suzuki K. Effectiveness of biofield therapy for individuals with sickle cell disease in Africa. Altern Ther Health Med. 2014 Jan-Feb;20(1):20-6. PMID 24445353
- See also: MOA International Corporation — http://www.moainternational.or.jp